CLINICAL TRIAL: NCT02881216
Title: Procedural Advantages of a Novel Drug-Eluting Coronary Stent With Ultra-Thin Struts and Bioabsorbable Abluminal Polymer Coating in an All-Comers Registry
Brief Title: Procedural Advantages of a Novel Drug-Eluting Coronary Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Haitham Abu Sharar, Principal Investigator, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Synergy Stent
Record Dates: First submitted 2016-08-15; First posted 2016-08-26 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- Common DES (Other): Group of Patients with narrowed coronary artery disease, who were treated with an implantation of currently established drug-eluting stents (Xience Prime, Promus Element plus, Resolute Integrity).
  Interventions: Device: Currently common drug-eluting stent (DES)
- Synergy Stent (Other): Group of Patients with narrowed coronary artery disease, who were treated with Synergy stent implantation
  Interventions: Device: Synergy Stent

INTERVENTIONS:
Device: Synergy Stent — Patients with narrowed coronary artery disease qualifying for PCI were treated with Synergy stent implantation.
  Other Names: Synergy Coronary Stent
  Arms: Synergy Stent
Device: Currently common drug-eluting stent (DES) — Patients with narrowed coronary artery disease qualifying for PCI were treated with DES implantation (Xience Prime, Resolute Integrity, Promus Element Plus)
  Other Names: DES including Xience Prime, Resolute Integrity, Promus Element Plus.
  Arms: Common DES

SUMMARY:
This study sought to compare procedural performance of a new coronary stent generation, that is already available in Germany, with hitherto established current drug-eluting stents.

ELIGIBILITY:
Inclusion Criteria:

* CAD for PCI, consecutive patients

Exclusion Criteria:

* Age under 18
* Bare Metal Stents or Scaffolds

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
In-hospital major cardiac adverse events | One week post-procedure
  In-hospital major cardiac adverse events were collected up to one week after procedure throughout the in-patients stay